CLINICAL TRIAL: NCT04861649
Title: Metabonomics of Chronic Obstructive Pulmonary Disease and Fecal Microbial Transplantation in the Treatment of Malnutrition
Brief Title: Metabonomics of COPD and Transplanting of Faecal Bacteria in the Treatment of Its Malnutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Asclepius Meditec Inc. (Industry)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT for COPD
Record Dates: First submitted 2021-04-05; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Fecal Microbiota Transplantation
Keywords: fecal microbiota transplantation, COPD, dystrophy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect and mechanism of fecal microbiota transplantation on patients with COPD malnutrition (Experimental): During COPD stable period, nasal and intestinal tubes were placed and fecal bacteria were transplanted from healthy people (three transplants per course of treatment).
  200ml of bacterial liquid was transplanted for each course, containing 40g of bacterial volume, transplanted consecutively for 3 times, once a day)
  Interventions: Biological: fecal microbiota transplantation

INTERVENTIONS:
Biological: fecal microbiota transplantation — The nasointestinal tube was placed and the fecal bacteria of healthy people were transplanted with liquid fecal bacteria (three transplants per course of treatment).
  200ml of bacterial liquid was transplanted for each course, containing 40g of bacterial volume, transplanted consecutively for 3 times, once a day)

SUMMARY:
Oxidative stress can affect the balance of intestinal flora and intestinal structure of patients, resulting in intestinal flora disorder. Its bacterial metabolites stimulate the parasympathetic nerve, regulate insulin secretion and other metabolic pathways of patients through neuroendocrine regulation, resulting in abnormal energy metabolism of lipids and sugars in the digestive tract, and finally lead to malnutrition.We hypothesized that fecal bacteria transplantation could reconstruct the normal intestinal flora, restore the intestinal digestion and absorption function of chronic obstructive pulmonary disease（COPD）patients and improve the state of malnutrition.

DETAILED DESCRIPTION:
1. improve the COPD patients with malnutrition is the key to improve the digestion and absorption function of chronic obstructive pulmonary disease (COPD) is one of the world's third most common cause of death, is characterized by progressive airflow limited, mainly by the long-term exposure to tobacco smoke and other harmful air pollutants.

   It has been reported that 20%-71% of COPD patients suffer from malnutrition, and there is a negative correlation between BMI and prognosis.

   There is increasing evidence that patients with COPD with lower BMI or fat-free mass index are associated with poorer prognosis and impaired long-term survival.

   At present, nutrition supplements are mainly used to solve the problem of COPD malnutrition, including vitamins and minerals, essential amino acids and biological amino acids, anti-inflammatory omega-3, high fat and high carbohydrate, etc., while the causes of COPD malnutrition and the relationship between COPD and metabolism have not been paid attention to.

   Although there is evidence that there is no malnutrition nutritional support can improve the prognosis of patients with COPD, but exist in patients with malnutrition, due to impaired digestion and absorption, increase nutrition supply, prone to patients with abdominal distension, vomiting, and diarrhea.

   Therefore, in order to improve malnutrition in patients with COPD, it is necessary to improve digestion and absorption function in patients with COPD.
2. improve digestion and absorption function, first of all, correct the oxidative stress caused by intestinal flora disorder as part of the systemic oxidative stress response, copd patients with intestinal oxidative stress, oxidative stress result of active oxygen free radicals on colon epithelium mucosa layer of mucin, lead to the loss of protein, mucous layer thickness can be reduced to 50%, resulting in changes in the structure of intestinal tract; In addition, under the action of active oxygen free radicals, epithelial cells of the digestive tract, the close connection between protein oxidation lead to intestinal epithelial permeability enhancement, on the one hand, the intestinal toxins can after connection into the intestinal permeability increased cells, affect the digestion and absorption function of intestinal cells, on the other hand, the oxidative stress products into the lumen of blood, lead to bacterial flora disorder, further affect intestinal digestion and absorption of food.

   The common clinical manifestations of intestinal flora disorder are: mild abdominal distension, diarrhea, nausea, vomiting, water and electrolyte disturbance, hypoproteinemia, malnutrition, and even shock. Therefore, in order to improve intestinal digestion and absorption function, it is necessary to correct intestinal flora disorder caused by oxidative stress.
3. intestinal flora and the relationship between nutrition, immunity, metabolism, neuroendocrine, normal human intestinal bacteria number, up to about 1013 ~ 1014 microbes, equivalent to 10 times of the total number of human tissue cells and its metabolites other tissue cells function to human body impact, the total number of genes at the same time, the intestinal bacteria coding is about more than 100 times of the total number of human genes, some experts believe that intestinal flora is one of the normal function of the human body organ, the abnormal organs, inevitably affects the health of human body.

Intestinal flora by helping to break down food and absorb nutrition, synthesis of nutrients, metabolites indirectly stimulate the nerve endocrine effects such as the host's nutritional status: promote ingested B vitamins (B3, B5, B6, B12) and other micronutrients, help absorb minerals (calcium, magnesium and iron, etc.), regulating metabolism of glucose and lipid storage.

Synthesis of micronutrients such as vitamin K, B12, biotin, folic acid and pantothenates; By affecting the integrity of mucosal epithelium, it plays an immune defense role.

Intestinal flora disturbance is related to the formation of metabolic diseases such as obesity and diabetes in the host. Rachels study showed that intestinal flora disturbance in rats can increase the production of acetate, and feeding acetate to rats can promote the secretion of insulin in rats, the mechanism of which is realized by the activation of acetate through the parasympathetic nerve.

The production of acetate increases, and the stimulation intensity of parasympathetic nerve is enhanced, which promotes insulin secretion, and promotes ghrelin secretion by consuming glucose and reducing hypoglycemia, leading to obesity.

A recent study also showed that the intestinal microbiome shifted from lean donors to patients with metabolic syndrome, resulting in increased insulin sensitivity of the receptors.4) animal models and patients with copd, there exist dysbacteriosis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of COPD
2. Tobacco use: current or former smokers with a continuous smoking history of more than 1 year.
3. Subjects are willing and able to complete the follow-up according to the plan.
4. Subjects can cooperate to complete relevant examination items.
5. Compliance: Subjects must be willing to return to the hospital and complete all visits and evaluations according to the protocol.

Exclusion Criteria:

1. Having a significant disease or condition other than COPD that, in the Investigator's judgment, would put the subject at risk for participating in the study or affect the study outcome and the subject's ability to participate in the study.
2. Women who are pregnant or breastfeeding or who plan to become pregnant during the study period.
3. Digestive system: ① patients with known gastrointestinal organic diseases.

   ② Complicated with intestinal double infection, such as Clostridium difficile infection, EHEC, Salmonella, Shigella, Campylobacter, plague and cytomegalovirus;

   ③ patients with various acute infections, tumors, severe arrhythmias, mental disorders, drug or alcohol addiction; (4) pregnant or lactating women; (5) Use of antibiotics or probiotics within the last 4 weeks; (6) There are taboo witnesses for this study; (7) Clinical investigators who were conducting other related COPD studies at the time of enrollment or within 3 months before enrollment;
4. Complicated with serious primary diseases of heart, liver, kidney, hematopoietic system and other important organs or systems.
5. Patients with lower back, chest and abdomen injuries or after surgery.
6. People with mental disorder or cognitive impairment.
7. Non-compliance: Subjects did not follow the study procedures, including non-compliance to complete the journal.
8. Informed consent validity is in doubt: Subjects with a history of psychosis, mental retardation, poor motivation, substance abuse (including drugs and alcohol), or other medical conditions that limit the effectiveness of informed consent in this study.
9. Obesity (BMI≥28) Hyperlipidemia (1.5 times the upper limit of normal value of plasma total cholesterol > or 1.5 times the upper limit of normal value of triglyceride BBB>; Confirmed diabetic patients; Diagnosed cancer patients; Have used any antibiotics or antibiotics in the last 2 weeks.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes of intestinal flora in COPD malnutrition subjects during the whole 6 months | 6 months
  The changes of intestinal flora were detected by 16SrDNA technology during the 6 months.
Nutritional indicators in COPD malnutrition subjects during the whole 6 months | 6 months
  including prealbumin, nutritional risk screening 2002 and scored patient-generated subjective global assessment.
the changes of COPD | 6 months
  The number of acute exacerbations in the previous year and the time of the last acute exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Zeguang Zheng, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Yimeng Xv, Study Chair — The First Affiliated Hospital of Guangzhou Medical University; Peiyan Zhong, Study Chair — The First Affiliated Hospital of Guangzhou Medical University; Ni Liu, Study Chair — The First Affiliated Hospital of Guangzhou Medical University; Shixian Ye, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Fecal Microbiota Transplantation, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
the main evaluation index and the secondary evaluation index of all participants will be share in 3 months after the end of this study.